CLINICAL TRIAL: NCT06217796
Title: A Single-Center, Open Label, Phase 4 Study of the Safety and Efficacy of Fixed Combination Phenylephrine 2.5%-Tropicamide 1% Ophthalmic Solution (Mydcombi®) Administered With the Mydcombi Dispenser for Pupil Dilation (THE MIST-2.1 STUDY)
Brief Title: Safety and Efficacy of Fixed Combination Phenylephrine-Tropicamide for Pupil Dilation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eyenovia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EYN-MYD-TP-41PM
Record Dates: First submitted 2024-01-04; First posted 2024-01-22 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-02

CONDITIONS: Mydriasis
Keywords: Mydriasis
MeSH Terms: conditions — Mydriasis | interventions — Tropicamide

STUDY DESIGN:
Intervention Model Description: All subjects receive the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Open Label Treatment (Other): Single metered spray
  Interventions: Combination Product: MydCombi

INTERVENTIONS:
Combination Product: MydCombi — A single metered spray administered with the MydCombi dispenser
  Other Names: tropicamide and phenylephrine hydrochloride ophthalmic spray 1%/2.5%

SUMMARY:
Subjects will receive ½ of the approved dose of MydCombi to determine the dilation curve with the reduced dose.

DETAILED DESCRIPTION:
MydCombi is approved for inducing mydriasis for diagnostic procedures and in conditions where short term pupil dilation is desired. The approved dose is 1 metered spray to the cornea of each eye to be dilated to be repeated after 5 minutes. This study will define the dilation of the pupil with ½ of the approved dose - a single metered spray to the cornea of each eye.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide signed written consent prior to participation in any study-related procedures.
* Ability to return for the study treatment visit.
* Photopic screening pupil diameter ≤ 3.5 mm in each eye.
* Females not of childbearing potential or negative pregnancy test

Exclusion Criteria:

* Pregnant or Lactating
* Clinically significant abnormalities of the eye
* Active eye disease
* Using medication that can effect pupil dilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Bennett, MS, Study Director — Eyenovia Inc.
Locations (1):
- SUNY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Treatment: A single metered spray of Mydcombi (tropicamide and phenylephrine hydrochloride ophthalmic spray)1%/2.5%
Period: Overall Study
Arm/Group | Open Label Treatment
Started | 30
Completed | 30 (One subject was excluded from analysis due to not meeting inclusion/exclusion criteria)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects meeting inclusion/exclusion criteria
Groups:
- Open Label Treatment: Single metered spray of MydCombi
  MydCombi: A single metered spray administered with the MydCombi dispenser
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 36.4 [20 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject declined to provide race
  Participants
    number analyzed (Participants) | 28
    American Indian or Alaska Native | 0
    Asian | 9
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 7
    White | 11
    More than one race | 1
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
Iris Color [Count of Participants; unit: Participants]
  Blue Iris | 2
  Brown Iris | 26
  Green Iris | 1
  Hazel Iris | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Pupil Diameter
Description: Mean change in pupil diameter at 30 minutes from the time of drug dose versus baseline, as measured by digital pupillometry in highly photopic conditions
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 58
millimeters
  Change from Baseline | 3.73 (1.293)
  Pupil Diameter | 6.46 (1.411)

2. Secondary Outcome: 6.0 mm or Greater at 30 Minutes
Description: Percentage of eyes achieving pupil diameter of 6.0 mm or greater
Time Frame: 30 minutes
Measure: Number; unit: percentage of eyes >6.0 mm
Units Other Than Participants: Eyes
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 58
percentage of eyes >6.0 mm | 67.2

3. Secondary Outcome: 7.0 mm or Greater at 30 Minutes
Description: Percentage of eyes achieving pupil diameter of 7.0 mm or greater
Time Frame: 30 minutes
Measure: Number; unit: percentage of eyes >7.0 mm
Units Other Than Participants: Eyes
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 58
percentage of eyes >7.0 mm | 43.1

4. Secondary Outcome: Distribution of Pupil Diameters
Description: Distribution of pupil diameters at 15, 30, 60, 90, 150, 210 and 360 minutes
Time Frame: 360 minutes
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 58
millimeters
  Baseline | 2.73 (0.446)
  15 Minutes | 4.80 (1.335)
  30 Minutes | 6.46 (1.411)
  60 minutes | 6.95 (1.255)
  90 Minutes | 6.70 (1.249)
  150 Minutes | 6.09 (1.360)
  210 Minutes | 5.18 (1.334)
  360 Minutes | 3.51 (0.774)

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | Open Label Treatment
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Treatment (N=30)
Dry Eye (Eye disorders) | 1 (1)
Instillation Site Pain (Eye disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT06217796/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT06217796/SAP_001.pdf